CLINICAL TRIAL: NCT02211599
Title: Post-Prandial Substrate Utilization in Response to the Inclusion of Sweetened Beverage to Meals With Different Levels of Protein Content
Brief Title: Fat Burning After a Meal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: USDA Grand Forks Human Nutrition Research Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: GFHNRC507
Record Dates: First submitted 2014-08-05; First posted 2014-08-07 (Estimated); Last update posted 2022-02-02 (Actual); Status verified 2022-01

CONDITIONS: Postprandial Effect of Carbohydrate Beverage Consumption
Keywords: protein; carbohydrate; lipid; oxidation; fat; sugar; juice; obesity
MeSH Terms: conditions — Platelet Glycoprotein IV Deficiency; Obesity | interventions — Proteins; Sugar-Sweetened Beverages

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 15% protein meal and sweetened beverage (Experimental): Breakfast and lunch will each contain 15% protein. A sweetened flavored beverage will be served with each meal; one drink will be sweetened with sugar and the other with sucralose (a non-nutritive sweetener). Order will be randomized.
  Interventions: Other: 15% protein; Other: Sweetened beverage
- 30% protein meal and sweetened beverage (Experimental): Breakfast and lunch will each contain 30% protein. A sweetened flavored beverage will be served with each meal; one drink will be sweetened with sugar and the other with sucralose (a non-nutritive sweetener). Order will be randomized.
  Interventions: Other: 30% protein; Other: Sweetened beverage

INTERVENTIONS:
Other: 15% protein — Meal to provide 15%en from protein.
  Arms: 15% protein meal and sweetened beverage
Other: 30% protein — Meal to provide 30%en from protein.
  Arms: 30% protein meal and sweetened beverage
Other: Sweetened beverage — Beverage sweetened with either sugar (sucrose) or sucralose (non-nutritive sweetener).

SUMMARY:
The purpose of the study is to determine how adding a carbohydrate beverage to a meal with different protein levels affects the rate at which one's body burns fats, sugars, and proteins.

ELIGIBILITY:
Inclusion Criteria:

* BMI less than 25 kg/m2
* ability to sign the consent form
* availability of transportation

Exclusion Criteria:

* percent body fat greater than or equal to 25% for males and 35% for females
* allergies to any study foods
* more than a 10% change in body weight within the past 2 months
* current or planned pregnancy
* lactation
* metabolic illness/disease(s)
* active cancer or in short-term remission (less than 3 years)
* infectious diseases
* alcohol or drug abuse
* tobacco use
* presence of acute illness
* taking medications known to affect energy expenditure and appetite

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Postprandial lipid oxidation rate | 4 hours after meal consumption

SECONDARY OUTCOMES:
Energy expenditure measured by postprandial thermogenesis | 4 hours after meal consumption
Postprandial protein oxidation | 4 hours after meal consumption
Postprandial carbohydrate oxidation | 4 hours after meal consumption

CONTACTS AND LOCATIONS:
Overall Officials: Shanon Casperson, PhD, Principal Investigator — USDA Grand Forks Human Nutrition Research Center; James Roemmich, PhD, Principal Investigator — USDA Grand Forks Human Nutrition Research Center
Locations (1):
- USDA Grand Forks Human Nutrition Research Center, Grand Forks, North Dakota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Casperson SL, Hall C, Roemmich JN. Postprandial energy metabolism and substrate oxidation in response to the inclusion of a sugar- or non-nutritive sweetened beverage with meals differing in protein content. BMC Nutr. 2017 Jul 21;3:49. doi: 10.1186/s40795-017-0170-2. eCollection 2017. PMID 32153829